CLINICAL TRIAL: NCT03123601
Title: Feasibility of Risk Sign Displays to Prevent Falls, Dehydration and Pulmonary Aspiration in Nursing Homes: a Clinical Study Protocol
Brief Title: Feasibility of Risk Sign Displays to Prevent Falls, Dehydration and Pulmonary Aspiration in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Neurológico Sénior (Other)
Collaborators: University of Lisbon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CNS2017-01
Record Dates: First submitted 2017-03-07; First posted 2017-04-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Nursing Home Residents
Keywords: Nursing home; Falls; Dysphasia; Choking; Dehydration
MeSH Terms: conditions — Aphasia; Airway Obstruction; Dehydration

STUDY DESIGN:
Intervention Model Description: All patients, with chronic neurologic diseases selected from a nursing home, will be invited to participate. At baseline patients will undertake a screening risk assessment and it will be attributed a correspondent risk display. Study duration will be a minimum of 3 months per participant, including daily record of events and monthly interview assessments. Events data will be compared with historical data extracted retrospectively from medical and nursing charts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Risk sign displays (Experimental): At baseline patients will undertake a screening risk assessment and it will be attributed a correspondent risk display. Study duration will be a minimum of 3 months per participant, including daily record of events and monthly interview assessments. Events data will be compared with historical data extracted retrospectively from medical and nursing charts.
  Interventions: Device: Risk sign displays

INTERVENTIONS:
Device: Risk sign displays — Set of sign displays designed to communicate fall, dehydration and pulmonary aspiration risks and reflect on tailored interventions to manage these events in nursing homes. Risk sign displays are:
  * Small, lightweight rubber coloured bracelets with phrases related with the different risks: "prevent rather than fall", "contain to protect", "drink to hydrate" and "avoid choking".
  * Small and coloured signposts next to head of patients bed that are believed to offer some key advantages and increase technically the quality of immediate communication of information and data regarding procedures. It is expected to have greater subject compliance once they will have discrete messages with thoughtful design and colour.

SUMMARY:
BACKGROUND: Prior research has shown a relationship between dehydration, falls and pulmonary aspiration among older adults in nursing and health care facilities, which contributes to its loss of independence and quality-of-life. Is believed that improving communication among health professional decreases the number of adverse events in institutionalized patients. This study will evaluate the feasibility of a set of sign displays designed to communicate fall, dehydration and pulmonary aspiration risks and will reflect on tailored interventions to manage these events in nursing homes.

METHODS AND ANALYSIS: This will be a national, single-center, feasibility study. All patients, with chronic neurologic diseases selected from a nursing home, will be invited to participate. At baseline patients will undertake a screening risk assessment and it will be attributed a correspondent risk display. Study duration will be a minimum of 3 months per participant, including daily record of events and monthly interview assessments. Events data will be compared with historical data extracted retrospectively from medical and nursing charts.

DETAILED DESCRIPTION:
1. Preparation phase - teaching session for health professionals An initial teaching session will be held to train and familiarize health professionals with the usage of the sign displays and corresponding intervention procedures. The training will also consist of memorizing/training the definition given to falls, dehydration and pulmonary aspiration and redefining registration of such events in the software. During the training session, any queries from the professionals will be explained. The investigators expect the training will last 60 minutes. This training will be accompanied by written information with the definition of a fall, pulmonary aspiration and dehydration, and specific instructions on what procedures to undertake for each risk sign display. Additionally, the researcher will exemplify the procedure practically, if needed.
2. Screening All patients will be invited to participate if they fulfil inclusion criteria. The nurse team from CNS nursing home will propose patients for recruitment and a multidisciplinary team will discuss and decided their study inclusion. In case of incapacity for the patients to give informed consent, family members will then be asked for consent and authorization of screening visit. Informed consent containing comprehensive information about objectives, duration, procedures, voluntariness and possible risks of study participation, will be obtained from patients before any study related proceedings. During the screening visit, an explanation of the objective and compliance needed for the study will be given to the participants and caregivers and all questions will be considered and answered.

   Demographics data, clinical manifestations and disease management, co-morbidities and past medical conditions will be obtained using a structured questionnaire. Also a brief clinical assessment of risk of falling, pulmonary aspiration and dehydration will be done.

   In the end of screening and risk assessment, the correspond risk displays will be given to patient by the investigator.

   2.1) Clinical Scales

   Mini Mental State Examination (MMSE) The Mini Mental State Examination is a brief 30-point questionnaire that is used to quantitatively assess cognition. The MMSE test includes simple questions and problems in a number of areas: the time and place of the test, repeating list of words, arithmetic, language use and comprehension, and copying a drawing. It can be used to screen for cognition impairment, to estimate the severity of cognitive impairment at a given point in time, to follow the course of cognitive changes in an individual over time, and to document an individual's response to treatment.

   Time Up and Go (TUG) Time Up and Go is a quick capacity measure to for functional mobility and a good predictor of subject's ability to independently walk outside safely. This clinical test is recommended by MDS review of measurement Instruments to assess posture, gait, and balance in Parkinson's disease and in the latest physiotherapy guidelines to Parkinson's disease. In this test is asked to participant to get up from a standard chair, walk 3m at a comfortable and safe speed and then turn walk to back to sit in the chair.

   Morse Falls Scale The Morse fall scale assesses the risk of falling for hospital in-patients or those in long-term care, in particular evaluates: falls history, the presence of comorbidities, the use of walking aids, mental status and whether or not patients are on intravenous therapy.

   Swallowing Disturbance Questionnaire (SDQ) The Swallowing Disturbance Questionnaire (SDQ) for PD patients is a validated self-reporting 15-item questionnaire on swallowing disturbances that appear in the oral and pharyngeal phases of swallowing. Fourteen questions rated by a four-point scale (0 for no disturbance and 3 for severe disturbance), and one ''yes/no'' question (yes was scored 2.5 and no was scored 0.5).

   GULP Dehydration Risk Screening Tool The GULP is a screening tool to assess geriatric dehydration risk. It includes a score from 0 to 7 points for three categories (24 h fluid intake; urine colour; clinical risk factors for dehydration). Based on results, the GULP tool recommends an hydration management plan, engaging like this the patient in self-monitoring of urine and verbal prompts.
3. Diary Record In the end of each nursing shift all events of falls, near falls, dehydration and pulmonary aspiration will be recorded in documents specifically created for that purpose by the working staff of CNS.
4. Monthly Visits At the end of each month, an interview will be performed to patients and a self-completed questionnaire will be handed to health professionals. Both will be questioned regarding overall acceptability levels and asked for any encountered problems regarding the use of the displays. Additionally, these moments will include questions on clarity of the instructions, reminder of the event definitions and the registration procedures.

   Importantly, investigators recognize that the visit interview is not flawless, because participants may have forgotten some of their complaints by the time of the visit interview. To their knowledge, there is no study that has previously studied whether recall interviews must be made weekly or whether more-frequent visits would be sufficient to obtain a reliable estimate of information. For this study, a monthly period was considered reasonable and particularly more helpful and feasible in future large trials with long follow-up periods.

   All visit interviews will be performed by the investigator and will take no more than 10 minutes.
5. Monthly reports In the end of each month, as strategy to keep health professionals informed and to remember the importance of registering, a newsletter will be sent to all CNS staff. This will contain information about the study duration and will present a summary of the number of participants in the study (number of patients recruited and number of drop-outs) and of the event recorded in that month.
6. Data collection of events It will also collect, in relation to all CNS residents, historical data related to falls, dehydration and pulmonary aspiration events retrospectively from medical and nursing chats within the period of the study and the same period, one year before.

ELIGIBILITY:
Inclusion criteria:

* Male or female staying at CNS nursing home for long term care;
* Risk of falling and/or dysphagia and/or dehydration defined by brief screening assessment;
* Being interested in participating in this study;
* Signing an informed consent form;
* Willing to comply with the monthly interviews required
* Eligibility validated by CNS health professionals in the multidisciplinary clinical meeting

Exclusion criteria:

* Having significant active psychiatric problems (example: hallucinations, confusion, psychosis) that aggravates patient´s symptoms when dealing with the use of sign displays;
* Inability participate according to the CNS health professionals' judgement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Patients' adherence trough the number of times and reasons to taken off the risk display or refused to use during the period of the study and/or withdrawing from the study | Minimum of 3 months

SECONDARY OUTCOMES:
Patients' satisfaction with the sign displays measured with a 7-point likert scale and open-ended questions. | Minimum of 3 months
Health professionals' satisfaction measured with sign displays through 7-point likert scale and open-ended questions regarding the overall benefits of using the displays and overall perception of its impact on decreasing risk. | Minimum of 3 months
Comparison to historical medical and nursing charts data review of the relative frequency of number of events per number of days of hospitalization registered during the period of the study, with in an equal period of time, one year before. | Minimum of 3 months
Type and frequency of adverse events recorded during the period of the study | Minimum of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim J Ferreira, MD, PhD, Principal Investigator — Campus Neurológico Sénior
Locations (1):
- Campus Neurológico Sénior, Torres Vedras, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duarte M, Bouca-Machado R, Domingos J, Godinho C, Ferreira JJ; CNS risk prompt display study group. Feasibility of using risk prompts to prevent falls, dehydration and pulmonary aspiration in nursing homes: a clinical study protocol. Pilot Feasibility Stud. 2018 Jan 25;4:39. doi: 10.1186/s40814-018-0236-1. eCollection 2018. PMID 29416872